CLINICAL TRIAL: NCT05570058
Title: A Multi-Cohort, Randomised, Placebo-Controlled Phase 2a Study to Assess the Safety, Pharmacokinetics, Pharmacodynamics and Clinical Activity of Ascending Doses of RXC007 in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: Assess the Safety, Pharmacokinetics, Pharmacodynamics and Clinical Activity of RXC007 in Idiopathic Pulmonary Fibrosis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Redx Pharma Ltd (Industry)
Collaborators: Simbec-Orion Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: RXC007/0002
Record Dates: First submitted 2022-09-28; First posted 2022-10-06 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: IPF; Fibrosis
Keywords: Lung; Respiratory; Fibrosis; IPF
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 (Experimental): 12:4 (RXC007 : Placebo) Dose level 1: 12 weeks (84 days) dosing
  Interventions: Drug: RXC007; Drug: Placebo
- Cohort 2 (Experimental): 12:4 (RXC007 : Placebo) Dose level 2: 12 weeks (84 days) dosing
  Interventions: Drug: RXC007; Drug: Placebo
- Expansion Cohort (Experimental): 12:4 (RXC007 : Placebo) Dose level 3: 12 weeks (84 days) dosing
  Interventions: Drug: RXC007; Drug: Placebo

INTERVENTIONS:
Drug: RXC007 — RXC007 will be administered in the form of oral capsules at 3 potential dose levels: 20 mg, 50mg and 70 mg in 5 cohorts. 12 patients of cohorts 1, 2 and the Expansion cohort will receive RXC007. The Dosage regimen is BID or QD.
Drug: Placebo — The placebo will be administered in the form of oral capsules at each dose level to 4 of the 16 participants within cohorts 1, 2 and the Expansion cohort. The Dosage regimen is BID or QD

SUMMARY:
The purpose of the study is to assess the safety and tolerability of RXC007 when given for 12 weeks (84 days), alone and in combination with nintedanib or pirfenidone.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the study drug RXC007.

The main objectives of this study are as follows:

* To determine the safety and tolerability (degree to which side effects of a drug can be tolerated) of RXC007 when it is administered as twice daily doses over a period of up to 12 weeks (84 days).
* To investigate the concentration of RXC007 (how much drug is in your blood), how this changes over a period of time and to evaluate whether there are differences in the concentration between different dose strengths of RXC007.
* To investigate the effect of RXC007 on the body (known as pharmacodynamics) by analysing the levels of certain biomarkers in the body and to assess the effect of RXC007 on markers associated with Idiopathic Pulmonary Fibrosis (IPF). Biomarkers are markers within the body such as a molecule or compound made by cells in the body, which can be measured and used to identify a particular disease.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥40 to 80 years at the time of signing the informed consent.
* Diagnosis of IPF within 5 years of Screening based on the modified ATS/ERS/JRS/ALAT IPF guidelines for diagnosis and management of IPF (Raghu et al, 2018) and confirmed on independent central imaging review.
* Combination of HRCT pattern, as assessed by central reviewers, consistent with diagnosis of IPF (see the modified ATS/ERS/JRS/ALAT IPF guidelines [Raghu et al, 2018]).
* FVC % predicted ≥50% predicted of normal at Screening, with no clinically significant deterioration between the Screening Visit and randomisation, as determined by the Investigator.
* DLco (Hb-adjusted) at screening ≥30%.
* In the main study, participants receiving treatment for IPF with nintedanib or pirfenidone are allowed if on treatment for at least 3 months and on a stable dose for at least 4 weeks prior to Screening and during Screening.
* In patients who are not on any treatment for IPF but have previously received nintedanib or pirfenidone, there needs to be a washout period ≥4 weeks prior to Screening.
* No clinically significant abnormalities, in the opinion of the investigator, in vital signs (e.g., blood pressure, pulse rate, respiration rate, oral temperature) within 28 days before first dose of IMP.

Exclusion Criteria:

* Currently receiving or planning to initiate treatment for IPF with agents not approved for that indication.
* FEV1/FVC ratio <0.7 at Screening, pre-bronchodilator use.
* Lower respiratory tract infection requiring antibiotics within 4 weeks of Screening or during Screening.

  4. The extent of emphysema in the lungs exceeds fibrosis, based on central review of HRCT scans.
* Need for continuous oxygen supplementation, defined as >15 hours/day.
* Acute IPF exacerbation within 6 months of Screening or during Screening.
* Clinical diagnosis of any connective-tissue disease (including, but not limited to, scleroderma, polymyositis/dermatomyositis, systemic lupus erythematosus, and rheumatoid arthritis) or a diagnosis of interstitial pneumonia with autoimmune features as determined by the Investigator applying the recent ERS/ATS research statement [Fischer et al 2015]. Note: Serological testing is not needed if not clinically indicated.
* Disease other than IPF with a life expectancy of less than 12 weeks.

Additional exclusion criteria for the Translational Science Sub Study

* Participants with any contra-indication to bronchoscopy and alveolar lavage including tracheal stenosis, pulmonary hypertension, severe hypoxia, or hypercapnia.
* Patients in the sub study are not permitted to receive nintedanib or pirfenidone within 3 weeks of randomisation and throughout the Treatment period. (Note: background IPF treatment should not be stopped for the purpose of eligibility)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2025-01-09 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of AEs and SAEs Changes in safety laboratory parameters, vital signs, and ECGs | From Day 1 to post-study follow up visit (12 weeks)
  The primary endpoints of the study include the incidence and severity of AEs and SAEs
Number of participants who report a change from normal range values for laboratory safety parameters (serum biochemistry, serum haematology or urinalysis) from first dose on Day 1 to post-study follow up visit. | From Day 1 to post-study follow up visit (12 weeks)
  This primary endpoint will report the number of participants within all cohorts of study who record a value which is deemed as outside of the normal range (regardless of clinical significance) for any of the serum biochemistry, serum haematology or urinalysis parameters as defined in the study protocol following first dose administration on Day 1 up to completion of the post-study visit
Number of participants who report a change from normal range values for vital signs parameters (blood pressure, pulse rate, respiration rate, oral body temperature) from first dose on Day 1 to 12 weeks of treatment | From Day 1 to post-study follow up visit (12 weeks)
  This primary endpoint will report the number of participants within all cohorts of the study who record a value which is deemed as outside of the normal range (regardless of clinical significance) for any of the vital signs parameters (systolic/diastolic blood pressure, pulse rate, respiration rate, oral body temperature) as defined in the study protocol following first dose administration on Day 1 up to completion of the post-study visit
Number of participants who report a change from normal range values for any of the associated 12-Lead ECG parameters (heart rate, QT interval and QTcF interval) from first dose on Day 1 up to completion of the post-study visit. | From Day 1 to post-study follow up visit (12 weeks)
  This primary endpoint will report the number of participants within all cohorts of the study who record a value which is deemed as outside of the normal range (regardless of clinical significance) for any of the 12-Lead ECG parameters (heart rate, QT interval and QTcF interval) as defined in the study protocol following first dose administration on Day 1 up to 12 weeks of treatment

SECONDARY OUTCOMES:
Pharmacokinetic Parameters - Maximum plasma concentration (Cmax) | For Cycle1 Day1 pre-dose, 1, 2, 3, 4, 8 h post-dose. For Cycle1 Day8 pre-dose, 1, 2, 3, 4, 8 h post-dose for all BID schedules. If the schedule is changed to QD, for Cycle1 Day8 will include a 24 h post-dose sample (Cycle1 Day9). On Cycle2 Day1 pre-dose.
  Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for RXC007. This endpoint will report the summary of derived pharmacokinetic parameters for the maximum observed concentration (Cmax) of RXC007 in plasma for all cohorts.
Minimum observed plasma concentration (Cmin) | For Cycle1 Day1 pre-dose, 1, 2, 3, 4, 8 h post-dose. For Cycle1 Day8 pre-dose, 1, 2, 3, 4, 8 h post-dose for all BID schedules. If the schedule is changed to QD, for Cycle1 Day8 will include a 24 h post-dose sample (Cycle1 Day9). On Cycle2 Day1 pre-dose.
  Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for RXC007. This endpoint will report the summary of derived pharmacokinetic parameters for the minimum observed concentration (Cmin) of RXC007 in plasma for all cohorts.
Pharmacokinetic Parameters - Time to maximum observed concentration (Tmax) | For Cycle1 Day1 pre-dose, 1, 2, 3, 4, 8 h post-dose. For Cycle1 Day8 pre-dose, 1, 2, 3, 4, 8 h post-dose for all BID schedules. If the schedule is changed to QD, for Cycle1 Day8 will include a 24 h post-dose sample (Cycle1 Day9). On Cycle2 Day1 pre-dose.
  Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for RXC007. This endpoint will report the summary of derived pharmacokinetic parameters for the time to maximum observed concentration (Tmax) of RXC007 in plasma for all cohorts.
Pharmacokinetic Parameters - Terminal elimination half-life (t1/2) | For Cycle1 Day1 pre-dose, 1, 2, 3, 4, 8 h post-dose. For Cycle1 Day8 pre-dose, 1, 2, 3, 4, 8 h post-dose for all BID schedules. If the schedule is changed to QD, for Cycle1 Day8 will include a 24 h post-dose sample (Cycle1 Day9). On Cycle2 Day1 pre-dose.
  Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for RXC007. This endpoint will report the summary of derived pharmacokinetic parameters for the terminal elimination half-life (t1/2) of RXC007 in plasma for all cohorts
Pharmacokinetic Parameters - Elimination rate constant (λz) | For Cycle1 Day1 pre-dose, 1, 2, 3, 4, 8 h post-dose. For Cycle1 Day8 pre-dose, 1, 2, 3, 4, 8 h post-dose for all BID schedules. If the schedule is changed to QD, for Cycle1 Day8 will include a 24 h post-dose sample (Cycle1 Day9). On Cycle2 Day1 pre-dose.
  Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for RXC007. This endpoint will report the summary of derived pharmacokinetic parameters for the elimination rate constant (λz) of RXC007 in plasma for all cohorts.
Pharmacokinetic Parameters - Area under the concentration-time curve (AUC) extrapolated to infinity (AUC0-inf) | For Cycle1 Day1 pre-dose, 1, 2, 3, 4, 8 h post-dose. For Cycle1 Day8 pre-dose, 1, 2, 3, 4, 8 h post-dose for all BID schedules. If the schedule is changed to QD, for Cycle1 Day8 will include a 24 h post-dose sample (Cycle1 Day9). On Cycle2 Day1 pre-dose.
  Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for RXC007. This endpoint will report the summary of derived pharmacokinetic parameters for the area under the concentration-time curve (AUC) extrapolated to infinity (AUC0-inf) of RXC007 in plasma for all cohorts.
Pharmacokinetic Parameters - Total apparent clearance following extravascular administration (CL/F) | For Cycle1 Day1 pre-dose, 1, 2, 3, 4, 8 h post-dose. For Cycle1 Day8 pre-dose, 1, 2, 3, 4, 8 h post-dose for all BID schedules. If the schedule is changed to QD, for Cycle1 Day8 will include a 24 h post-dose sample (Cycle1 Day9). On Cycle2 Day1 pre-dose.
  Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for RXC007. This endpoint will report the summary of derived pharmacokinetic parameters for the total apparent clearance following extravascular administration (CL/F) of RXC007 in plasma for all cohorts.
Pharmacokinetic Parameters - Apparent volume of distribution following extravascular administration (Vz/F) | For Cycle1 Day1 pre-dose, 1, 2, 3, 4, 8 h post-dose. For Cycle1 Day8 pre-dose, 1, 2, 3, 4, 8 h post-dose for all BID schedules. If the schedule is changed to QD, for Cycle1 Day8 will include a 24 h post-dose sample (Cycle1 Day9). On Cycle2 Day1 pre-dose.
  Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for RXC007. This endpoint will report the summary of derived pharmacokinetic parameters for the apparent volume of distribution following extravascular administration (Vz/F) of RXC007 in plasma for all cohorts.
Pharmacokinetic Parameters - Area under the plasma concentration-time curve during a dosing interval at steady state (AUCss) | For Cycle1 Day1 pre-dose, 1, 2, 3, 4, 8 h post-dose. For Cycle1 Day8 pre-dose, 1, 2, 3, 4, 8 h post-dose for all BID schedules. If the schedule is changed to QD, for Cycle1 Day8 will include a 24 h post-dose sample (Cycle1 Day9). On Cycle2 Day1 pre-dose.
  Plasma samples will be obtained in order to evaluate defined plasma pharmacokinetic parameters for RXC007. This endpoint will report the summary of derived pharmacokinetic parameters for the area under the concentration-time curve (AUC) at steady state of RXC007 in plasma for all cohorts.
% predicted and absolute volume change from baseline in Forced Vital Capacity (FVC) at 12 weeks [central review] | At Screening (Day28 to Day-1), Cycle1 Day1 pre-dose and post-dose, Cycle1 Day8, Cycle1 Day15, Cycle1 Day22, Cycle2 Day1(The day after Cycle1 Day28), Cycle2 Day15, Cycle3 Day1, Cycle3 Day28, End Of Treatment: last day of the dosing Day 21
  Information on Forced Vital Capacity (FVC) for the 6 months prior to study entry will be collected. Spirometry testing (without bronchodilator use) will be performed at all scheduled study visits in clinic. For each patient, spirometry testing should be conducted at approximately the same time of day.
% predicted and absolute change from baseline in carbon monoxide diffusion capacity (DLCO) | At Screening (day28 to Day-1), Cycle1 Day1 pre-dose, Cycle1 Day15, Cycle2 Day1 (The day after Cycle1 Day28)
  Carbon monoxide diffusion capacity will be measured in clinic

CONTACTS AND LOCATIONS:
Overall Officials: Philip Molyneaux, MD, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust; Toby Maher, MD, Principal Investigator — University of Southern California, USA
Locations (31):
- Medical University of Vienna, Vienna, Austria
- Belgium (2):
  - E PNE UZ Leuven, Leuven
  - CHU De Liège, Liège
- Pneumologicka klinika 1.LF UK a, Prague, Czechia
- Italy (8):
  - Azienda Ospedaliero-Universitaria "Ospedali-Riuniti" di Ancona, Ancona
  - Azienda Ospedaliero Universitaria Policlinico ''G.Rodolico-San Marco'', Catania
  - Colonello D'avanzo Hospital, Foggia
  - PO Vito Fazzi, Lecce
  - Ospedale S. Giuseppe Milano, Milan
  - Azienda Ospedaliera Universitaria of Modena, Modena
  - Fondazione Policlinico Universitario A. Gemelli, Roma
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Poland (3):
  - University Clinical Centre in Gdansk, Gdansk
  - Barlicki University Hospital, Lodz
  - Institute of Tuberculosis and Lung Diseases in Warsaw, Warsaw
- Spain (7):
  - Policlinica Barcelona, Barcelona
  - Hospital Universitario Clínic de Barcelona, Barcelona
  - L'Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela
- University Hospital of Geneve, Geneva, Switzerland
- United Kingdom (8):
  - Belfast City Hospital, Belfast
  - Queen Elizabeth Hospital, Birmingham
  - Royal Papworth Hospital NHSFT, Cambridge
  - Royal Infirmary of Edinburgh, Edinburgh
  - Guy's Hospital, London
  - Royal Brompton Hospital, London
  - Altnagelvin Area Hospital, Londonderry
  - Churchill Hospital, Oxford University Hospitals NHS Trust, Oxford

IPD SHARING:
Plan to Share IPD: No
At this stage, it is not planned that any IPD information will be shared with other researchers outside of the Sponsor and Clinical Research Organisation undertaking the conduct of this study.